CLINICAL TRIAL: NCT04237181
Title: Results of FilmArray® Gastro-intestinal Panel (GI Panel) and Serum Procalcitonin (PCT) in Acute Colitis and Infectious Diarrhea in the Emergency Department.
Brief Title: Results of FilmArray® Gastro-intestinal Panel and Serum Procalcitonin in Acute Colitis and Infectious Diarrhea in the ER
Acronym: PRODIARRAY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Biofire (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP191050; 2019-A02924-53 (Other: ANSM)
Record Dates: First submitted 2020-01-17; First posted 2020-01-23 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Acute Diarrhea; Acute Colitis of Presumed Infectious Origin
Keywords: Infectious Diarrhea; Colitis; PCR multiplex; PCT
MeSH Terms: conditions — Dysentery; Colitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acute diarrhoea or colitis presumed to be of infectious origin (Other)
  Interventions: Device: Filmarray PCR multiplex-PCT assay

INTERVENTIONS:
Device: Filmarray PCR multiplex-PCT assay — Filmarray PCR multiplex gastro intestinal panel on stools and serum PCT dosage

SUMMARY:
Acute diarrhea and acute colitis of infectious origin are common reasons for consultation at the emergency department. The current etiological diagnostic approach is limited to the determination of markers of inflammation, such as CRP and blood leukocytes, which lack specificity and sensitivity for bacterial infection. The stool culture can detect bacterial pathogens in the stool with a result at least 48 hours later and a positivity rate <50%.

This study will describe the procalcitonin (PCT) concentrations (a biomarker of bacterial infection) in this population to evaluate its usefulness depending on the viral or bacterial etiology identified by stool multiplex gastro-intestinal PCR panel (GI panel) and stool culture.

The investigators hypothesize that PCT levels will be higher if the GI panel or the stool culture identifies a bacteria or a parasite, as it is the case in respiratory tract infections. If there is a detection of a virus by the GI panel or both the stool culture and the GI panel are negative, the investigators expect that PCT values will be lower or negative.

the investigators will include the patients admitted to the ED with a suspicion of infectious diarrhea or acute colitis in order to have a large representative panel of infectious diarrhea etiologies.

Only the patients having a blood sample prescribed as the routine care will be included. The blood sample is useful for dosing CRP and whole blood cell count (WBC), which are part of current biologic analyses performed in this context. After getting the patient's consent, the investigator will add the PCT dosage in blood sampling and will ask the patient to provide a stool sample, in order to have a stool culture and to perform an extended investigation for the pathogens through multiplex PCR technology (Filmarray ®GI panel).

The physician will be asked if all these results (the ones ordered currently together with the dosage of PCT and the GI panel) will change his/her decision to start an antibiotic.

Patients will receive a phone call at day 15 after their initial admission in the emergency department and will be asked if he/she has consulted a new physician or if a new treatment by antibiotics was started.

Data collection procedures: Data from the medical file will be collected by the investigators and the emergency department clinical research assistant. All the data will be pseudonymized. The collection will be done at the day of admission in the emergency department and after the phone interview at Day15.

DETAILED DESCRIPTION:
Acute diarrhea and acute colitis of infectious origin are common reasons for consultation at the emergency department. The current etiological diagnostic approach is limited to the determination of markers of inflammation, such as CRP and blood leukocytes, which lack specificity and sensitivity for bacterial infection. The stool culture can detect bacterial pathogens in the stool with a result at least 48 hours later and a positivity rate <50%.

This study will describe the procalcitonin (PCT) concentrations (a biomarker of bacterial infection) in this population to evaluate its usefulness depending on the viral or bacterial etiology identified by stool multiplex gastro-intestinal PCR panel (GI panel) and stool culture.

The investigators hypothesize that PCT levels will be higher if the GI panel or the stool culture identifies a bacteria or a parasite, as it is the case in respiratory tract infections. If there is a detection of a virus by the GI panel or both the stool culture and the GI panel are negative, the investigators expect that PCT values will be lower or negative.

The investigators will include the patients admitted to the ED with a suspicion of infectious diarrhea or acute colitis in order to have a large representative panel of infectious diarrhea etiologies.

Only the patients having a blood sample prescribed as the routine care will be included. The blood sample is useful for dosing CRP and whole blood cell count (WBC), which are part of current biologic analyses performed in this context. After getting the patient's consent, the investigator will add the PCT dosage in blood sampling and will ask the patient to provide a stool sample, in order to have a stool culture and to perform an extended investigation for the pathogens through multiplex PCR technology (Filmarray ®GI panel).

The physician will be asked if all these results (the ones ordered currently together with the dosage of PCT and the GI panel) will change his/her decision to start an antibiotic.

Patients will receive a phone call at day 15 after their initial admission in the emergency department and will be asked if he/she has consulted a new physician or if a new treatment by antibiotics was started.

Data collection procedures: Data from the medical file will be collected by the investigators and the emergency department clinical research assistant. All the data will be pseudonymized. The collection will be done at the day of admission in the emergency department and after the phone interview at Day15.

Statistical justification for sample size: This will be a pilot study to describe the results of PCT concentration and multiplex GI panel. As to our knowledge, there is no published study reporting PCT concentrations in this population. This preclude a sample, size calculation. The investigators will include as much patients as possible during one year in order to cover the epidemiological seasonal variations and to obtain a convenient sample of at least 100 patients.

Statistical methods description: Clinical and biological data will be reported as median and interquartile range or mean +/- SD. PCT values will be reported as median and IQR, respectively if a there is a viral infection, a documented infection (bacterium or parasite) or no pathogen identified by GI panel and/or stool culture (bacteria). Patient's characteristics and PCT results will be compared in all groups, using as a reference, the group where no pathogen is observed. A sub-group analysis will be performed on colitis and acute diarrhea respectively, to find out if there is any difference with the variables analyzed as both pathologies are not managed in the same way.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for patients presenting an acute diarrhoea :

1. Patients over 18 years of age,
2. Signed informed consent form
3. Having a social security insurance,
4. Attending the emergency department for Acute diarrhoea (at least three loose or liquid stools a day for less than 15 days)
5. For whom a blood test in the emergency department is ordered as a standard of care

Inclusion criteria for patients presenting an infectious colitis :

1. Patients over 18 years of age,
2. Signed informed consent form
3. Having a social security insurance,
4. Attending the emergency department for a documented colitis presumed to be of infectious origin, for whom a blood test in the emergency department is planned, defined by:

   1. at least one of the following symptoms: abdominal pain, fever, diarrhoea and
   2. Elevated white blood cell count (> 10.000/mm3) or CRP (> 10 mg/l) and
   3. An abdominal CT scan showing a thickening of at least segmental colonic walls.

Exclusion Criteria:

1. Recent abdominal surgery of less than one month
2. Pregnancy
3. Inflammatory bowel disease
4. Patients under curatorship or guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2020-03-24 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
PCT concentration according to each type of pathogens identified using GI panel and stool cultures (bacteria, virus, parasites). | Day 1
  The median PCT concentration will be reported in the three main etiological group (viruses, bacteria, parasites) identified by stool culture and GI panel

SECONDARY OUTCOMES:
Positivity rate and distribution of pathogens identified by the GI panel and stool culture | Day 1
  Positivity Rate of GI Panel and stool culture given in percentage (%) and the distribution of pathogens found if positive, divided in 3 groups (virus, bacteria and parasites)
Rate of antibiotic therapy initiated in the ER and in the first following 15 days | Day 1 and 15
  Rate of antibiotics use given in percentage (%)
Number of days of antibiotic exposure at day 15 | Day 15
  Number of days on antibiotics for each patient
Rate of antibiotics prescription before and after results of the GI panel and PCT (Day 1) | Day 1
  Rate (%) of intention to start an antibiotic before the results of the GI panel and rate (%) of antibiotic's prescription after the results of the GI panel and PCT

CONTACTS AND LOCATIONS:
Locations (1):
- Pitié Salpetriere, Paris, France

IPD SHARING:
Plan to Share IPD: No